CLINICAL TRIAL: NCT07059819
Title: Evaluation of Local Hyperthermia for the Treatment of Cervical Intraepithelial Neoplasias 3 Months After Treatment: a Multicenter, Single-blind, Randomized Controlled Trial
Brief Title: Local Hyperthermia for the Treatment of Cervical Persistent High-risk Infection
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Gao Xinghua, Professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HH20241031
Record Dates: First submitted 2025-03-26; First posted 2025-07-11 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-10

CONDITIONS: Cervical Intraepithelial Neoplasia (CIN); Human Papillovirus
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Hyperthermia (Experimental)
  Interventions: Device: Local hyperthermia device
- Placebo (Placebo Comparator)
  Interventions: Device: Local hyperthermia device

INTERVENTIONS:
Device: Local hyperthermia device — Local hyperthermia at 44℃ for 30 mins on cervical region, at days of 1,2,3 and 17, 18.

SUMMARY:
Human papillomavirus(HPV) infect epithelial cells and have the capacity to stimulate cell abnormal hyperplasia, especially by those high-risk HPV types. HPV vaccine primarily targeting HPV6/11/16/18 has been available and makes it possible to prevent cervical cancer. However, a large population was left unvaccinated, specifically for those aged ones. In clinic, patients harboring high-risk HPV is quite prevalent in China or other developing nations. Removing the virus and prevention of malignant transformation is required.

Mild local Hyperthermia with a certain temperature range has been successfully used in the treatment of some diseases. It has been utilized in the treatment of some neoplasm, fungal and HPV infections. Investigators' study found that local hyperthermia at 44°C could cleared HPV in more than half of the patients with HR-HPV in cervical area. So the purpose of the study is to evaluate the effective of local hyperthermia in the treatment of cervical intraepithelial neoplasias grade I and II after 3 months. Appropriate control arms were designed for different conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old; generally healthy gynecological conditions, normal sexual life; high risk HPV for persistent at least 3 months; Cervical biopsy CIN or no cytological changes; signed informed consent

Exclusion Criteria:

* Pregnant woman; local or systematic treatment within 3 months; Comorbidity of other severe gynecological inflammation, infection, or tumor; Comorbidity of other serious illnesses; no guarantee of timely treatment and follow-up.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Clearance of high-risk HPV | 3 and 6 months after treatment
  Detection of HPV genotype by PCR (21 subtypes)

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China